CLINICAL TRIAL: NCT04586140
Title: Operation of the Groupe Hospitalier Paris Saint-Joseph Clinical Ethical Reflection Assistance Group During the COVID-19
Brief Title: Operation of the GHPSJ Clinical Ethical Reflection Assistance Group During the COVID-19 Period
Acronym: ETHICOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ETHICOVID
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Ethics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID-19 infection: This study will be carried out on patient data usually collected as part of their care. The patients were infected with COVID-19 and hospitalized between 03/25/2020 and 05/07/2020, and who benefited from GAREC's intervention.
- Nursing staff AND GAREC Members: This study also concerns data collected in the context of semi-structured interviews with health professionals, in a prospective manner. These are caregivers who are members of GARED or who called on GAREC between 25/03/2020 and 07/05/2020.

SUMMARY:
Between March and May 2020, Ile-de-France hospitals faced an influx of patients infected with the COVID 19 virus. Faced with the scale of the pandemic, the aggressiveness of this pathology, severe respiratory complications and the shortage of resuscitation beds , the teams had to make difficult decisions on the therapeutic strategy, the orientation of patients in the event of respiratory distress and their intensive care status. To do this, each establishment reflected in an emergency context on procedures for collegial deliberation and assistance in ethical reflection, based on the recommendations of the National Consultative Ethics Committee and learned societies such as the French Society. of Anesthesia and Resuscitation or the French Society of Support and Palliative Care.

Some hospitals had already institutionalized the ethical approach upstream of the health crisis. For example, the Groupe d'Aide à la Réflexion Éthique Clinique (GAREC) was created in November 2005 within the Paris Saint-Joseph Hospital Group. GAREC is a collegial and multidisciplinary entity, made up of 8 members who intervene at the request of caregivers when a clinical situation turns out to be ethically complex. He gives an advisory opinion, the decision belonging to the referring physician.

At the start of the COVID period, GAREC changed its structure, organization and operation in order to respond to the multiple issues posed by the complexity of the health situation.

This study seeks to analyze the adaptation mechanisms put in place by this group during the epidemic period as well as the nature of the benefit provided to the caregivers who requested it, to the patients and to their relatives.

* Adaptation mechanisms: during the COVID period, GAREC was extended to other paramedical professions (psychologists, nurses), thus increasing from 8 to 15 members. It has set up 2 weekly meetings, an on-call duty and on-call duty. The requests were made easier: they could be done by phone, by email, day or night. Several questions emerge: What were the motivations for enlarging the group? How were the members integrated into this group? What were its operating methods? How and by whom was it seized? For what purpose? Were the intervention teams multidisciplinary?
* Nature of the benefit provided by GAREC: it will be approached by semi-structured interviews via a qualitative research method.

This work is part of a broader reflective perspective:

* What representation of ethics underlies this device?
* Does the institutionalization of ethics help to enhance or make invisible what ethics owes to daily healthcare practices?
* To what extent does the institutionalization of clinical ethics make health institutions more human and virtuous?
* Under what conditions can a device like GAREC go beyond the role of ethical guarantor and transform the institution and nursing practices in the service of a collective reflective approach? This study will be carried out on patient data usually collected as part of their care and on data collected through semi-structured interviews with healthcare professionals. As such, it fits into the perspective of grounded theory.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Major
  * Hospitalized for a COVID-19 infection and for which GAREC intervened between 03/25/20 and 05/07/20
* Caregivers:

  * GAREC members (between 8 and 15 caregivers)
  * Having called on GAREC (between 10 and 20 caregivers)

Exclusion Criteria:

* Patients

  * Patient under guardianship or curatorship
  * Patient deprived of liberty
  * Patient under legal protection
  * Patient objecting to the use of their data for this research
* Caregivers o Caregiver opposing the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for COVID-19 infection who benefited from GAREC's intervention between 03/25/2020 and 05/07/2020.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Interest of GAREC | Year 1
  This outcome is to evaluate the benefit of nursing staff in the ethical process. In a qualitative study like this, no primary endpoint is established.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Lorraine de WARREN, Nurse, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- See also: Related Info — https://www.coreb.infectiologie.com/UserFiles/File/procedures/rpmo-ethique-rea-covid-19-vf-24-corr26-mar20-2.pdf